CLINICAL TRIAL: NCT01160679
Title: Effectiveness of Atypical Antipsychotics on Anhedonic Features in Patients With Schizophrenia
Acronym: PLEASURE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Marketing Company Medical Director, AstraZeneca
Other Study IDs: NIS-NKR-SER-2010/1
Record Dates: First submitted 2010-07-07; First posted 2010-07-12 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Schizophrenia
Keywords: anhedonic features in patients with schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, multi-center, 12 weeks naturalistic NIS trial will be conducted in 25 hospitals in naturalistic treatment setting. There will be no experimental component associated with this study and all observational activities have to be part of routine care visit: baseline (week 0), week 4 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis of schizophrenia meeting the Diagnostic and Statistical Manual of Mental Disorders,(DSM-IV-TR) criteria
* Patients who already take one atypical at inclusion it is started at least 1 week and up to 4 weeks before the inclusion

Exclusion Criteria:

* Meeting the criteria for any other (than schizophrenia) DSM-IV Axis I
* Patients with antipsychotic combinations (more than two agents)
* Patients who are already on any mood stabilizers and antidepressant
* Known lack of response to clozapine or treatment with clozapine within 4 weeks prior to enrollment
* Patients who have been treated with antipsychotics in depot formulations for the last two months
* Previous enrollment or randomisation of treatment in the present NIS
* Patients who had participated in other clinical trials within 4 weeks prior to enrollment period
* Pregnant women or women who are breast-feeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of psychiatry of 25 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The change of total score of SHAPS | At baseline
The change of total score of SHAPS | At 12 weeks

SECONDARY OUTCOMES:
Changes of Clinical Global Impression (CGI)-Severity score | At baseline
Changes of Clinical Global Impression (CGI)-Severity score | At 12 weeks
Proportion of patients having a score of 1 or 2 in CGI-I score | At 12 weeks
Proportion of significantly improved patients in SHAPS total score (more than 30%) | At baseline
The mean change MADRS total score | At baseline
The mean change MADRS total score | At 12 weeks
Proportion of significantly improved patients in SHAPS total score (more than 30%) | At 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Woo Han, MD, PhD, Study Chair — Department of Psychiatry
Locations (12):
- South Korea (12):
  - Research Site, Busan, Busan
  - Research Site, Gongju, Chungcheongnam-do
  - Research Site, Daegu, Daegu
  - Research Site, Daejeon, Daejeon
  - Research Site, Chuncheon, Gangwon-do
  - Research Site, Anyang-si, Gyeonggi-do
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Yongin-si, Gyeonggi-do
  - Research Site, Gyeongju, Gyeongsangbuk-do
  - Research Site, Changnyeong, Gyeongsangnam-do
  - Research Site, Seoul, Seoul